CLINICAL TRIAL: NCT00005947
Title: A Randomized, Double Blind, Placebo Controlled Trial of Immunotherapy With Autologous Antigen-Loaded Dendritic Cells (Provenge) for Asymptomatic Metastatic Hormome-Refractory Prostate Cancer
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Elizabeth Smith, Dendreon Corporation
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9901 CDR0000067868; DEN-D9901; NCI-G00-1789
Record Dates: First submitted 2000-07-05; First posted 2004-03-05 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- sipuleucel-T (Active Comparator)
  Interventions: Biological: sipuleucel-T
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: sipuleucel-T — Autologous peripheral blood mononuclear cells, including antigen presenting cells, that have been activated in vitro with a recombinant fusion protein, PAP-GM-CSF. Treatment consist of 3 doses administered approximately 2 weeks apart.
  Other Names: APC8015, Provenge
  Arms: sipuleucel-T
Biological: Placebo — Approximately one-third of the autologous quiescent antigen presenting cells (APCs) prepared from a single leukapheresis procedure. A course of therapy consists of 3 complete doses given at approximately 2-week intervals.
  Arms: Placebo

SUMMARY:
Rationale: Vaccines may make the body build an immune response to kill tumor cells. It is not yet known if vaccine therapy is effective for prostate cancer.

Purpose: Randomized phase III trial to determine the effectiveness of vaccine therapy in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
Objectives:

I. Compare the time to progression, time to development of disease-related pain, and incidence of grade 3 or worse treatment-related adverse events in patients with asymptomatic metastatic hormone refractory adenocarcinoma of the prostate treated with APC8015 versus control infusion. II. Compare response rate and duration of response in these patients.

Outline: This is a randomized study. Patients are randomized to one of two treatment arms. Arm I: Autologous dendritic cell precursors (ADCP) are harvested on weeks 0, 2, and 4. Patients receive APC8015 comprised of ADCP activated with prostatic acid phosphatase-sargramostim (GM-CSF) fusion protein IV over 30 minutes beginning 2 days after each harvest for a total of 3 infusions. Arm II: ADCP are harvested as in arm I. Patients receive unactivated ADCP IV over 30 minutes beginning 2 days after each harvest for a total of 3 infusions. Pain is assessed weekly for up to 3 years or until 4 weeks after objective disease progression. Patients are followed monthly for up to 3 years or until disease progression. At the time of disease progression, patients treated on arm II may receive treatment on Protocol D9903.

Projected Accrual: A total of 120 patients (80 in arm I and 40 in arm II) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria include:

* Metastatic disease as evidenced by soft tissue and/or bony metastases.
* Baseline PSA value of at least 5 ng/mL. All subjects must have stable or rising PSA.
* Tumor progression after hormonal therapy.
* Hormonal therapy consisting of castration by orchiectomy or LHRH agonists for treatment of prostate cancer. Castration levels of testosterone (< 50 ng/dL) must be documented for all subjects including subjects who underwent orchiectomy as therapy for cancer of the prostate.
* A subject is eligible if he initially responded to antiandrogen withdrawal (> 25% decrease in PSA) but at the time of registration demonstrated tumor progression. A subject is eligible if he failed to respond to antiandrogen withdrawal.
* Subjects have no cancer-related pain and do not regularly require analgesics for cancer-related pain.
* ECOG Performance Status of 0 or 1.
* Life expectancy of at least 16 weeks.
* Adequate hematologic, renal, and liver function.

Exclusion Criteria include:

* Visceral organ metastases (e.g., liver, lung, brain) or cytologically positive effusions (e.g., pleural effusions or ascites).
* Metastatic disease expected to be in need of radiation therapy within 4 months.
* Concurrent therapy with experimental agents.
* Systemic corticosteroids at doses greater than 40 mg hydrocortisone per day for any reason other than treatment of prostate cancer within the previous 6 months without prior approval.

Please note that there are additional eligibility criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 1999-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Small, MD, Study Chair — University of California, San Francisco
Locations (34):
- United States (34):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Office of Glenn Tisman, Whittier, California
  - Office of Barry S. Berman, Orlando, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Albany Regional Cancer Center, Albany, New York
  - Center for Medical Oncology, Garden City, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - St. Luke's-Roosevelt Hospital, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - AKSM Clinical Research Corporation, Columbus, Ohio
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Abington Hematology Oncology Associates, Incorporated, Abington, Pennsylvania
  - Bryn Mawr Urology, Bryn Mawr, Pennsylvania
  - Office of Guy Bernstein, M.D., Bryn Mawr, Pennsylvania
  - Saint Mary Regional Cancer Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Hematology/Oncology Associates of NE Pennsylvania, P.C., Scranton, Pennsylvania
  - American Oncology Resources, Dallas, Texas
  - Devine Tidewater Urology, Norfolk, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Hematology Oncology Northwest, P.C., Tacoma, Washington

REFERENCES:
- [Background] Higano CS, Schellhammer PF, Small EJ, Burch PA, Nemunaitis J, Yuh L, Provost N, Frohlich MW. Integrated data from 2 randomized, double-blind, placebo-controlled, phase 3 trials of active cellular immunotherapy with sipuleucel-T in advanced prostate cancer. Cancer. 2009 Aug 15;115(16):3670-9. doi: 10.1002/cncr.24429. PMID 19536890
- [Result] Small EJ, Schellhammer PF, Higano CS, Redfern CH, Nemunaitis JJ, Valone FH, Verjee SS, Jones LA, Hershberg RM. Placebo-controlled phase III trial of immunologic therapy with sipuleucel-T (APC8015) in patients with metastatic, asymptomatic hormone refractory prostate cancer. J Clin Oncol. 2006 Jul 1;24(19):3089-94. doi: 10.1200/JCO.2005.04.5252. PMID 16809734
- [Derived] Ju M, Fan J, Zou Y, Yu M, Jiang L, Wei Q, Bi J, Hu B, Guan Q, Song X, Dong M, Wang L, Yu L, Wang Y, Kang H, Xin W, Zhao L. Computational Recognition of a Regulatory T-cell-specific Signature With Potential Implications in Prognosis, Immunotherapy, and Therapeutic Resistance of Prostate Cancer. Front Immunol. 2022 Jun 23;13:807840. doi: 10.3389/fimmu.2022.807840. eCollection 2022. PMID 35812443
- [Derived] Small EJ, Higano CS, Kantoff PW, Whitmore JB, Frohlich MW, Petrylak DP. Time to disease-related pain and first opioid use in patients with metastatic castration-resistant prostate cancer treated with sipuleucel-T. Prostate Cancer Prostatic Dis. 2014 Sep;17(3):259-64. doi: 10.1038/pcan.2014.21. Epub 2014 Jun 24. PMID 24957547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between January 2000 and September 2004 across 16 clinical trial sites.
Pre-assignment Details: Participants were screened for evaluation of subject eligibility and performance of baseline tests/procedures.
Groups:
- Sipuleucel-T: All subjects randomized to receive sipuleucel-T.
  Autologous peripheral blood mononuclear cells, including antigen presenting cells, that have been activated in vitro with a recombinant fusion protein, PAP-GM-CSF. Treatment consist of 3 doses administered approximately 2 weeks apart.
- Placebo: All subjects randomized to receive placebo.
  Approximately one-third of the autologous quiescent APCs prepared from a single leukapheresis procedure. A course of therapy consists of 3 complete doses given at approximately 2-week intervals.
Period: Overall Study
Arm/Group | Sipuleucel-T | Placebo
Started | 82 | 45
Completed | 25 | 4
Not Completed | 57 | 41
Not completed — Death | 54 | 40
Not completed — Patient Refused to Continue | 2 | 1
Not completed — Site Closure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: All subjects randomized to receive placebo. Approximately one-third of the quiescent APCs prepared from a single leukapheresis procedure.
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T | Placebo | Total
Number analyzed (Participants) | 82 | 45 | 127
Age Continuous [Mean (Standard Deviation); unit: years] | 72.1 (8.1) | 71.1 (8.3) | 71.7 (8.1)
Age, Customized [Median (Full Range); unit: Years (Min, Max)] | 73.0 [47 to 85] | 71.0 [50 to 86] | 73.0 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 82 | 45 | 127

OUTCOME MEASURES:

1. Primary Outcome: Time to Objective Disease Progression
Description: The time to objective disease progression in patients with asymptomatic metastatic hormone-refractory prostate cancer treated with APC8015 (sipuleucel-T).
Time Frame: 36 months from randomization
Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Sipuleucel-T: All subjects randomized to receive sipuleucel-T.
- Placebo: All subjects randomized to receive placebo
Arm/Group | Sipuleucel-T | Placebo
Number analyzed (Participants) | 82 | 45
Weeks | 11.7 [9.1 to 16.6] | 10.0 [8.7 to 13.1]
Statistical Analysis 1: Comparison: Sipuleucel-T vs Placebo; Test type: Superiority or Other; p = 0.052, Log Rank; Hazard Ratio (HR) = 1.45, 95% CI [0.99 to 2.11] — Obtained from a Cox proportional hazards model with treatment group as the independent variable [placebo/sipuleucel-T]
Statistical Analysis 2: Comparison: Sipuleucel-T vs Placebo; Test type: Superiority or Other; p = 0.052, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.47 to 1.01] — Obtained from a Cox proportional hazards model with treatment group as the independent variable [sipuleucel-T/placebo]

2. Secondary Outcome: Overall Survival
Description: Overall Survival
Time Frame: From randomization to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sipuleucel-T | Placebo
Number analyzed (Participants) | 82 | 45
Months | 25.9 [20.0 to 32.4] | 21.4 [12.3 to 25.8]
Statistical Analysis 1: Comparison: Sipuleucel-T vs Placebo; ITT Population - all randomized participants; Test type: Superiority or Other; p = 0.010, Log Rank; Hazard Ratio (HR) = 1.71, 95% CI [1.13 to 2.58] — Cox proportional hazards model with treatment as the independent variable [placebo/sipuleucel-T]
Statistical Analysis 2: Comparison: Sipuleucel-T vs Placebo; ITT Population - all randomized participants; Test type: Superiority or Other; p = 0.010, Log Rank; Hazard Ratio (HR) = 0.586, 95% CI 2-sided [0.388 to 0.884] — Cox proportional hazards model with treatment as the independent variable [sipuleucel-T/placebo]

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Arm/Group | Sipuleucel-T | Placebo
Serious Adverse Events (participants affected / at risk) | 22/82 | 8/45
Other Adverse Events (participants affected / at risk) | 82/82 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (N=82) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bladder Obstruction (Renal and urinary disorders) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Heart rate irregular (Investigations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (N=82) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Constipation (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 12 | 5
Vomiting (Gastrointestinal disorders) | 10 | 1
Asthenia (General disorders) | 9 | 1
Chills (General disorders) | 51 | 4
Fatigue (General disorders) | 36 | 17
Feeling cold (General disorders) | 8 | 1
Influenza like illness (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 6 | 5
Pain (General disorders) | 5 | 5
Pyrexia (General disorders) | 28 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Weight decreased (Investigations) | 6 | 2
Anorexia (Metabolism and nutrition disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 10
Chest wall pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Shoulder pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Headache (Nervous system disorders) | 14 | 1
Paraesthesia (Nervous system disorders) | 13 | 2
Tremor (Nervous system disorders) | 8 | 0
Insomnia (Psychiatric disorders) | 1 | 4
Dysuria (Renal and urinary disorders) | 2 | 4
Haematuria (Renal and urinary disorders) | 5 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 4
Urinary retention (Renal and urinary disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Flushing (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A provision provides for sponsor review up to 45 days with the right to request modification based on disclosure of confidential information; extendable by 60 days to file a patent application.